CLINICAL TRIAL: NCT02509949
Title: Effects of Dexmedetomidine on Delirium After Living Donor Renal Transplantation in Adult Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, Tao Zhang, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DDRT
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Delirium After Living Donor Renal Transplantation
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine ivpump 0.2ug/kg/h during living donor renal transplantation.
  Interventions: Drug: Dexmedetomidine
- Saline (Placebo Comparator): Saline ivpump 0.2ug/kg/h during living donor renal transplantation.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Saline
  Arms: Saline

SUMMARY:
Delirium, an acute change in mental status, is a serious medical complication among hospitalized patients. Syndrome of delirium involves agitation, sleep disturbance, affective disorders and cognitive disruptions.

One vulnerable period for developing delirium is in the postoperative days. Postoperative delirium often initiates a cascade of adverse consequences including an increase in length of stay and hospital costs, and greater mortality. The investigators have observed that the incidence of postoperative delirium in patients after renal transplantation is about 20-30% in our hospital.

Several studies have revealed that dexmedetomidine, as a widely used sedative during anesthesia, can decrease the incidence of postoperative delirium after cardiac surgery. The investigators aim to examine whether administration of dexmedetomidine can reduce postoperative delirium after living donor renal transplantation in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 17 and < 60 years;
* American Society of Anesthesiology (ASA) I-III;
* admitted for living donor renal transplantation.

Exclusion Criteria:

* Patients with a history of drug abuse;
* preoperative history of schizophrenia, epilepsy, parkinsonism, use of cholinesterase inhibitor, inability to communicate in the preoperative period (coma, profound dementia, or language barrier).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium | Postoperative day 1-7.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China